CLINICAL TRIAL: NCT07206433
Title: Identification and Perceptions of Spoken Language Abilities After Transient Ischaemic Attack (TIA): An Exploratory, Longitudinal Study
Brief Title: Transient Ischemic Attack (TIA) and Spoken Language
Status: Not yet recruiting | Type: Observational
Sponsor: Newcastle University (Other)
Collaborators: Northumbria Healthcare NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: TIASPEECHPROTOCOL3132025
Record Dates: First submitted 2025-04-23; First posted 2025-10-03 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-04

CONDITIONS: TIA (Transient Ischemic Attack)
Keywords: TIA; Transient Ischemic Attack; speech; language
MeSH Terms: conditions — Ischemic Attack, Transient; Speech; Language

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Transient Ischaemic Attack (also known as TIA or 'mini-stroke') affects about 46,000 people in the UK each year. It is assumed that people recover fully within 24 hours. However, subtle problems with speaking, and confidence with their communication skills can be long-term. This project will be the first in depth exploration of speaking abilities after recent TIA where there seemed to be a full recovery.

The researchers will look for 90 volunteers for detailed testing. Thirty people who have had a TIA for the first time. For comparisons, the researchers will also include 60 volunteers without TIA (30 treated to prevent TIA and stroke; 30 who do not receive prevention treatments).

Aims and methods:

1. To find out if TIA makes speaking difficult.

   People will complete speaking tasks in a quiet place. For example, people will be asked to tell us about their weekend, what they think about climate change.
2. To find out if people are concerned about their speech and other thinking skills after TIA.

   People will fill in questionnaires to help us look into these issues.
3. To find out if speaking abilities and people's own views of their communication change over time (about three months after the TIA).

Discovering new knowledge about spoken communication after a TIA diagnosis could change the course of TIA research and care across health professions (speech-language therapy, psychology, audiology, neurology). Future studies could use speaking tasks to scrutinise further the complexity of subtle communication problems after TIA and determine which individuals are likely to have these problems. The project will raise understanding of these issues, enabling affected individuals to seek professional support. Finally, it will also guide development of new TIA recommendations and treatments for these problems thus improving people's quality of life.

DETAILED DESCRIPTION:
Montreal Cognitive Assessment (MoCA; (Nasreddine et al., 2005): Assesses general cognitive function; reliable and valid; different versions for repeated assessment (e.g., sentence repetition "I only know that John is the one to help today"; You'll hear a list of numbers and I'd like you to repeat them in the order you heard them).

Everyday Memory Questionnaire (Sunderland et al., 1986): Self-reported measure of cognitive skills many of which are about communication, language and reading (Likert scale) (e.g., forgetting the names of friends or relatives or calling them by the wrong names; getting lost or turning in the wrong direction on a journey or walk you have often been on).

Data analyses

For aims 1 and 2, the methods of analysis for each of the outcome measures is detailed below and will be in conducted in R.

Descriptive statistics by subgroup (medians, range, inter-quartile range) will be generated for each outcome measure (speech-related [primary, secondary], Everyday Memory Questionnaire, Communication Confidence Rating Scale for Aphasia).

Kruskal-Wallis non-parametric analysis of variance will be carried out for each outcome measure (alpha level .05). Post-hoc pairwise comparisons (using Dunn's test correction for multiple comparisons) for statistically significant results. Effect sizes will also be obtained.

Communication Confidence Rating Scale for Aphasia (Cherney et al., 2011): Self-reported confidence in communication activities (Likert scale) (e.g., how confident are you about your ability to talk with people? How confident are you that people understand you when you talk?)

Connected speech assessment tasks (Whitworth et al., 2015): Assesses connected speech skills, (e.g., can you tell me what you did last weekend? Can you remember a recent celebration such as a birthday, anniversary, wedding or party that you have been to? Can you tell me about it? What do you think about global warming and why?)

For aim 3, descriptive statistics (as above) will be generated for each outcome measure non-parametric Wilcoxon tests (alpha level 0.5) will be used. Effect sizes will also be obtained. These analyses will also be carried out in R.

ELIGIBILITY:
Inclusion Criteria: People aged 40-85 with a diagnosis of a single carotid circulation TIA.

Exclusion Criteria:

Younger than 40 years or older than 85 years of age.

English as a secondary language.

Neurological conditions affecting cognitive function (e.g., Parkinson's disease, dementia, stroke).

Self-reported, pre-existing speech or cognitive problems, developmental or acquired.

Demonstrate noticeable difficulties carrying out project-related tasks.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: TIA group: Individuals who have had a recent single medically confirmed TIA following an in-person review at a TIA clinic.
  Vascular risk factor group: People aged 40-75 with vascular risk factors (e.g., hypertension, diabetes, hyperlipidemia) who receive medical treatment for these conditions and have attended a TIA clinic but were not diagnosed with a TIA.
  Healthy group: People aged 40-75 who have no self-reported vascular risk factors for which they take medication.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Speech rate | From enrollment
  measured as number of words per minute
Mean length of sentence | From enrollment
  measured in number of words
Sentence complexity | From enrollment
  measured as number of complex sentences
Functional Memory Questionnaire | From enrollment
  Patient-reported measure of perceptions of memory, attention, language abilities;
  score range 0 to 140; higher scores mean a worse outcome
Communication Confidence Rating Scale for Aphasia | From enrollment
  Patient-reported measure of confidence of communication abilities;
  score range 0 to 600; higher scores mean worse outcome

SECONDARY OUTCOMES:
Filled pause rate | From enrollment
  Number of filled paused (i.e., "um" "uh", "ehm") over total number of words
Lexical richness | From enrollment
  measured as number of unique words over total number of words
Propositional idea density | From enrollment
  using the Computerized Propositional Idea Density Rater - CPIDER3 - Brown et al. (2008)

CONTACTS AND LOCATIONS:
Overall Officials: Christos Salis, PhD, Principal Investigator — Newcastle University; Lisa Shaw, MD, Study Chair — Newcastle University; Christopher Price, MD, Study Chair — Newcastle University; Mahmoud Kargar, MSc, Study Chair — Newcastle University
Locations (1):
- Newcastle University, Newcastle upon Tyne, Tyne and Wear, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided